CLINICAL TRIAL: NCT05083195
Title: The Effect of Individualized Home-Based Telerehabilitation Intervention on Physical Parameters and Activities of Daily Living in Individuals With Stroke
Brief Title: The Effect of Home-Based Telerehabilitation in Individuals With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Recep Ormen, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC-2021/62
Record Dates: First submitted 2021-10-08; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Stroke
Keywords: Telerehabilitation; Home-based; Physiotherapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): This group will perform their exercises with pre-prepared personalized exercise videos over the telerehabilitation system 3 times a week for 8 weeks.
  Interventions: Other: Home-based Telerehabilitation
- Control Group (Experimental): This group will perform exercises with personalized exercise brochures defined over the telerehabilitation system 3 times a week for 8 weeks.
  Interventions: Other: Exercise Brochure

INTERVENTIONS:
Other: Home-based Telerehabilitation — Balance, walking, strengthening exercise videos etc. taken in different positions will be uploaded to the telerehabilitation system. A personalized exercise program will be created from these exercises. This program will be defined to the account of the patient and the follow-up of the person will be carried out through the system.
  Arms: Telerehabilitation Group
Other: Exercise Brochure — Photos and explanations of exercises taken in different positions such as balance, walking, strengthening etc. will be uploaded to the telerehabilitation system. A personalized exercise brochure will be created from these exercises. This program will be defined for the patient's account and the patient will be asked to follow the exercises with this brochure.
  Arms: Control Group

SUMMARY:
Stroke is a clinical picture that develops due to occlusion or rupture of cerebral vessels and results in loss of cerebral functions. Stroke individuals face some limitations in managing daily activities such as walking, dressing, feeding and showering. Personal, environmental, and societal limitations have led to the development of new treatment strategies, such as telerehabilitation(TR), to meet the needs of stroke individuals and their caregivers.

In this study, patients will be randomized and divided into 2 groups in order to examine the effects of two different TR methods on physical parameters and activities of daily living in stroke patients. Baseline assessments will be made for both groups to determine functionality, activities of daily living, fall activity, quality of life, and level of fatigue. For 8 weeks, the TR group will do their exercises with exercise videos prepared on the system 3 times a week. The control group, on the other hand, will do their exercises with exercise brochures on the system 3 times a week for 8 weeks. After 8 weeks, assessments will be repeated. With telerehabilitation to be applied to individuals with stroke, it is aimed to increase functional capacity, independence in daily living activities and quality of life, and reduce the number of falls and fatigue levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stroke at least 1 year ago by a neurologist
* Modified Rankin score ≤3
* Have an internet infrastructure that can be accessed at home
* Not participated in a standardized physiotherapy program in the past 3 months

Exclusion Criteria:

* Presence of blurred or low vision problems
* Hearing and speech impairment at a level that will affect participation in the system
* Epilepsy
* Presence of pregnancy
* Having any cognitive problems that prevent using the system

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-08-04 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Single Leg Stance Test (The change between the initial value and the value after 2 months will be evaluated) | Baseline and end of weeks 8
  It is a functional assessment test that measures the patient's standing balance on one leg. It is applied for both legs of the patient with eyes open and closed.
Five Times Sit to Stand Test (The change between the initial value and the value after 2 months will be evaluated) | Baseline and end of weeks 8
  This test assesses functional lower extremity strength, transfer, balance, and fall risk. The time the patient sits and stands up from the chair 5 times is recorded.
Romberg Test (The change between the initial value and the value after 2 months will be evaluated) | Baseline and end of weeks 8
  The patient's standing time is recorded in an upright position with her feet open at shoulder level and arms free at the side of the body, with her eyes open and then closed, without losing her balance.
Independent Standing test (The change between the initial value and the value after 2 months will be evaluated) | Baseline and end of weeks 8
  It tests the patient's ability to stand in an upright position without any support or assistance, with her feet shoulder-width apart and arms free at the side of the body.
Katz Index of Independence in Activities of Daily Living (The change between the initial value and the value after 2 months will be evaluated) | Baseline and end of weeks 8
  It is a scale that measures the patient's ability to perform activities of daily living independently and evaluates the functional status.

SECONDARY OUTCOMES:
Modified Falls Efficacy Scale (The change between the initial value and the value after 2 months will be evaluated) | Baseline and end of weeks 8
  It is a 14-item scale that measures the patient's confidence in falling.
WHOQOL-BREF-TR (The change between the initial value and the value after 2 months will be evaluated) | Baseline and end of weeks 8
  It is a health-related quality of life scale developed by the World Health Organization. A national question was added to the Turkish version of the scale in addition to the original version.
Fatigue Severity Scale (The change between the initial value and the value after 2 months will be evaluated) | Baseline and end of weeks 8
  It is a scale that evaluates the severity of fatigue with 9 items that patients can answer on their own.
Global Rating of Change Scales | End of weeks 8
  It is a scale that evaluates how much the patient's current condition has changed compared to previous condition.
System Usability Scale | End of weeks 8
  It is a scale consisting of 10 questions widely used in the literature to evaluate the perceptibility and usability of interactive systems.

CONTACTS AND LOCATIONS:
Overall Officials: Recep Ormen, M.Sc, Principal Investigator — Istanbul University-Cerrahpasa Institute of Postgraduate Education; Yonca Zenginler Yazgan, PhD, Study Chair — Istanbul University-Cerrahpasa Faculty of Health Science
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakirkoy, Turkey (Türkiye)